CLINICAL TRIAL: NCT00255840
Title: "Safeguard the Household" - A Study of HIV Antiretroviral Therapy Treatment Strategies Appropriate for a Resource Poor Country
Brief Title: Evaluation of Two Anti-HIV Treatment Strategies in Resource-Limited South African Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CIPRA SA (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: James McIntyre, CIPRA SA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPRA-SA Project 1; U19AI053217 (NIH); 3U19AI053217-03S1 (NIH); 3U19AI053217-04S1 (NIH); 3U19AI053217-04 (NIH)
Record Dates: First submitted 2005-11-16; First posted 2005-11-21 (Estimated); Results first posted 2011-06-16 (Estimated); Last update posted 2011-06-21 (Estimated); Status verified 2011-06

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — efavirenz; Lamivudine; Lopinavir; Nevirapine; Stavudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Study-specified Antiretroviral regimen under care of HIV-trained medical doctor
  Interventions: Behavioral: Monitoring by an HIV-trained medical doctor; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Stavudine
- B (Active Comparator): Study-specified Antiretroviral regimen under care of HIV-trained primary care nurse
  Interventions: Behavioral: Monitoring by an HIV-trained primary care nurse; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nevirapine; Drug: Stavudine

INTERVENTIONS:
Behavioral: Monitoring by an HIV-trained medical doctor — Participants will receive care from an HIV-trained medical doctor
  Arms: A
Behavioral: Monitoring by an HIV-trained primary care nurse — Participants will receive care from an HIV-trained primary care nurse
  Arms: B
Drug: Efavirenz — 600 mg tablet taken orally daily
  Other Names: EFV
Drug: Lamivudine — 150 mg tablet taken orally daily
  Other Names: 3TC
Drug: Lopinavir/Ritonavir — 400 mg lopinavir/100mg ritonavir tablet taken orally twice daily
  Other Names: LPV/RTV
Drug: Nevirapine — 200 mg tablet taken orally for 14 days before taking a 200 mg tablet orally twice daily
  Other Names: NVP
Drug: Stavudine — Tablet taken orally daily. Dosage depends on weight.
  Other Names: d4T

SUMMARY:
The purpose of this study is to determine the effectiveness of several anti-HIV treatment strategies in resource-poor South African communities. The strategies being studied are using specially trained doctors or nurses to administer HIV care.

DETAILED DESCRIPTION:
The introduction of antiretroviral therapy (ART) for the treatment of HIV has dramatically improved morbidity and mortality for HIV infected people in the developed world. However, research data on the efficacy of ART regimens in developing countries, such as South Africa, are limited. There are an estimated 4.7 million HIV infected individuals in the South African population of about 40 million inhabitants. The greatest social impact may be achieved by treating an entire household affected by HIV to ensure maximum adherence to prescribed ART regimens and to minimize the sharing of antiretroviral drugs. This study will evaluate the effectiveness of ART given by an HIV-trained doctor compared to ART given by an HIV-trained primary health care nurse. Participants failing first-line therapy will receive a second-line regimen based on what medications are available at the clinic, with approval by the clinical safety team. Participants in this study will be recruited from resource-poor communities outside Johannesburg and Cape Town, South Africa.

This study will last 5 years. HIV infected people and other HIV infected members of their household 16 years of age and older will be enrolled. Study participants will receive first-line ART consisting of efavirenz (EFV) once daily, lamivudine (3TC) twice daily, and stavudine (d4T) twice daily. Women of childbearing potential who are unwilling to use acceptable forms of contraception and who have CD4 counts less than 250 cells/mm3 will receive 3TC twice daily; nevirapine (NVP) daily for 2 weeks, then twice daily; and d4T twice daily. Women who are pregnant at baseline, who become pregnant on study treatment, or who are unwilling to use acceptable methods of contraception and have CD4 counts of 250 cells/mm3 or more, or children who were previously exposed to NVP will receive 3TC twice daily, lopinavir/ritonavir (LPV/r) twice daily, and d4T twice daily. Participants will be randomly assigned to one of two arms. Arm 1 will receive ART under the monitoring care of an HIV-trained medical doctor, while Arm 2 will receive ART under the monitoring care of an HIV-trained primary health care nurse with training in HIV diagnosis and treatment. Participants who fail their first-line regimen will receive a second-line regimen but will remain in their treatment arms.

Study visits will occur at study entry; Weeks 2, 4, 8, and 12; and every 12 weeks thereafter. A physical exam, measurement of height and weight, tuberculosis (TB) and hepatitis B infection screening, blood collection, pill counts, and compliance/adherence and resource utilization counseling will occur at most visits. Participants will also be asked to complete quality of life and household cost questionnaires at selected visits. Study visits for participants who fail first-line treatment will occur at treatment failure, between Days 15 and 30, Week 4 post-treatment failure, every 4 weeks until Week 48 post-treatment failure, and every 12 weeks thereafter. A targeted physical exam, measurement of height and weight, TB infection screening, blood collection, pill counts, and compliance/adherence and resource utilization counseling will occur at most visits. Participants will also be asked to complete quality of life and household cost questionnaires at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Current severe CDC Category B AIDS-defining illness (with the exception of a single episode of bacterial sepsis or a single episode of zoster), OR history of a severe CDC Category B or C AIDS-defining illness, OR one CD4 count less than 350 cells/mm3 within 6 months prior to study entry
* Antiretroviral naive. A participant who previously received 6 weeks or less of post-exposure prophylaxis or short course therapy for the prevention of mother-to-child transmission are not excluded. More information on this criterion can be found in the protocol.
* Willing to use acceptable forms of contraception
* Parent or guardian willing to provide informed consent, if applicable

Exclusion Criteria:

* Current newly diagnosed CDC Category C AIDS-defining opportunistic infection or condition requiring acute therapy at the time of study entry. More information on this criterion can be found in the protocol.
* Therapy with agents with significant systemic myelosuppressive, neurotoxic, pancreatotoxic, hepatotoxic, or cytotoxic potential within 30 days prior to study entry
* Require certain medications
* Current alcohol or substance abuse that, in the opinion of the investigator, may interfere with the study
* Uncontrolled diarrhea (more than 6 stools per day for 7 consecutive days) within 30 days prior to study entry
* Diagnosis of or suspected acute hepatitis within 30 days prior to study entry
* Signs or symptoms of bilateral peripheral neuropathy of Grade 2 or greater at screening
* Inability to tolerate oral medication
* Any other clinical condition that, in the opinion of the investigator, may interfere with the study
* In the first trimester of pregnancy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 812 (Actual)
Dates: Start 2006-07; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James McIntyre, MBChB, MRCOG, Principal Investigator — Perinatal HIV Research Unit, Chris Hani Baragwanath Hospital; Ian Sanne, MBChB, Principal Investigator — University of the Witwatersrand, Thembaletu Clinic, Helen Joseph Hospital; Robin Wood, MBChB, FCP (SA), Principal Investigator — Department of Medicine, University of Cape Town

REFERENCES:
- [Background] Hosseinipour MC, Kazembe PN, Sanne IM, van der Horst CM. Challenges in delivering antiretroviral treatment in resource poor countries. AIDS. 2002;16 Suppl 4:S177-87. doi: 10.1097/00002030-200216004-00024. No abstract available. PMID 12699015
- [Background] Sanne I, van der Horst C. Research as a path to wide-scale implementation of antiretroviral therapy in Africa. J HIV Ther. 2004 Sep;9(3):65-8. PMID 15534564
- [Background] Wools-Kaloustian K, Kimaiyo S. Extending HIV care in resource-limited settings. Curr HIV/AIDS Rep. 2006 Nov;3(4):182-6. doi: 10.1007/s11904-006-0014-1. PMID 17032578
- [Derived] Brehm JH, Koontz DL, Wallis CL, Shutt KA, Sanne I, Wood R, McIntyre JA, Stevens WS, Sluis-Cremer N, Mellors JW; CIPRA-SA Project 1 Study Team. Frequent emergence of N348I in HIV-1 subtype C reverse transcriptase with failure of initial therapy reduces susceptibility to reverse-transcriptase inhibitors. Clin Infect Dis. 2012 Sep;55(5):737-45. doi: 10.1093/cid/cis501. Epub 2012 May 22. PMID 22618567
- [Derived] Orrell C, Cohen K, Conradie F, Zeinecker J, Ive P, Sanne I, Wood R. Efavirenz and rifampicin in the South African context: is there a need to dose-increase efavirenz with concurrent rifampicin therapy? Antivir Ther. 2011;16(4):527-34. doi: 10.3851/IMP1780. PMID 21685540
- [Derived] Sanne I, Orrell C, Fox MP, Conradie F, Ive P, Zeinecker J, Cornell M, Heiberg C, Ingram C, Panchia R, Rassool M, Gonin R, Stevens W, Truter H, Dehlinger M, van der Horst C, McIntyre J, Wood R; CIPRA-SA Study Team. Nurse versus doctor management of HIV-infected patients receiving antiretroviral therapy (CIPRA-SA): a randomised non-inferiority trial. Lancet. 2010 Jul 3;376(9734):33-40. doi: 10.1016/S0140-6736(10)60894-X. PMID 20557927

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-positive adult participants were recruited from February 2005 to December 2007 from two primary health care clinics, one in Masiphumelele, Cape Town and the other in Soweto, Johannesburg.
Groups:
- Antiretroviral Therapy Monitored by Medical Officer: First line antiretroviral regimen monitored by a HIV-trained medical doctor:
  1. Stavudine (>60 kg: 40 mg twice daily and <60 kg: 30 mg twice daily)
  2. Lamivudine (150mg twice daily) and
  3. Efavirenz (600mg daily). For women of child bearing potential with a CD4+ count <250 cells/mm3, Nevirapine (200 mg daily x 14 days, then 200 mg twice daily) and for women with a CD4+ count > 250 cells/mm3, Lopinavir/ritonavir (400/100mg twice daily).
- Antiretroviral Therapy Managed by Primary Health Care Nurse: First line antiretroviral regimen monitored by HIV-trained primary health care nurse:
  1. Stavudine (>60 kg: 40 mg twice daily and <60 kg: 30 mg twice daily)
  2. Lamivudine (150mg twice daily) and
  3. Efavirenz (600mg daily). For women of child bearing potential with a CD4+ count <250 cells/mm3, Nevirapine (200 mg daily x 14 days, then 200 mg twice daily) and for women with a CD4+ count > 250 cells/mm3, Lopinavir/ritonavir (400/100mg twice daily).
Period: Overall Study
Arm/Group | Antiretroviral Therapy Monitored by Medical Officer | Antiretroviral Therapy Managed by Primary Health Care Nurse
Started | 408 | 404
Completed | 345 | 334
Not Completed | 63 | 70
Not completed — Lost to Follow-up | 10 | 14
Not completed — Discontinued intervention | 53 | 56

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Antiretroviral Therapy Monitored by Medical Officer | Antiretroviral Therapy Managed by Primary Health Care Nurse | Total
Number analyzed (Participants) | 408 | 404 | 812
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 408 | 404 | 812
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.2612388 (7.1934154) | 32.9739630 (7.3921786) | 33.12 (7.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 276 | 297 | 573
  Male | 132 | 107 | 239
Region of Enrollment [Number; unit: participants]
  South Africa | 408 | 404 | 812

OUTCOME MEASURES:

1. Secondary Outcome: To Compare Subject Adherence to First Line Antiretroviral Treatment as Measured by Pill Count, Between the Two Primary Health Care Monitoring Models.
Time Frame: Throughout study
Reporting Status: Not Posted

2. Secondary Outcome: Drug Resistance HIV Mutations, Defined by Demonstration of Virologic Failure
Time Frame: Throughout the study
Reporting Status: Not Posted

3. Secondary Outcome: To Compare the Overall Clinical Safety of Antiretroviral Therapy, as Measured by the Occurrence of Clinical and Laboratory Grade 3 and 4 Adverse Events, Between Primary Health Care Monitoring Arms.
Time Frame: Throughout study
Reporting Status: Not Posted

4. Secondary Outcome: To Estimate the Total and Incremental Costs, From the Provider and Societal Perspectives, of the Two Approaches (the Primary Health Care Sister and Doctor) to the Provision of Antiretrovirals in Primary Health Care Services in Each Study Site.
Time Frame: Throughout study
Reporting Status: Not Posted

5. Primary Outcome: Cumulative Treatment Failure Rate of Participants on First Line Antiretroviral Therapy Monitored by Primary Health Care Nurses (Investigative Arm)is Not Inferior to the Cumulative Treatment Failure Rate of Participants Monitored by Doctors (Control Arm).
Description: Cumulative treatment failure is a composite endpoint made up of death, virological failure, toxicity failure and protocol-defined loss to follow-up failure.
Time Frame: 96 weeks
Population: The primary analysis was an intention-to-treat analysis of any treatment failure with use of Cox proportional hazards regression.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Antiretroviral Therapy Monitored by Medical Officer | Antiretroviral Therapy Managed by Primary Health Care Nurse
Number analyzed (Participants) | 408 | 404
Percentage of participants | 44 [39 to 49] | 48 [43 to 52]

ADVERSE EVENTS:
Arm/Group | Antiretroviral Therapy Monitored by Medical Officer | Antiretroviral Therapy Managed by Primary Health Care Nurse
Serious Adverse Events (participants affected / at risk) | 126/408 | 153/404
Other Adverse Events (participants affected / at risk) | 194/408 | 119/404
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antiretroviral Therapy Monitored by Medical Officer (N=408) | Antiretroviral Therapy Managed by Primary Health Care Nurse (N=404)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Leucopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 7 (7)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastrointestinal symptoms NOS (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 1 (1)
Right Upper Quadrant Pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Hyphema (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Rectal Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ruptured Appendix (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death (General disorders) | 3 (3) | 1 (1)
Swelling of Legs (General disorders) | 1 (1) | 0 (0)
Weakness (General disorders) | 1 (1) | 1 (1)
Adverse Drug Reaction (General disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 1 (2)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2) | 0 (0)
Immune Reconstitution Syndrome (Immune system disorders) | 1 (1) | 0 (0)
Abcess (Infections and infestations) | 0 (0) | 3 (4)
Bronchopneumonia (Infections and infestations) | 1 (1) | 0 (0)
Buboes (Infections and infestations) | 1 (1) | 0 (0)
Cerebral Toxoplasmosis (Infections and infestations) | 1 (1) | 0 (0)
Chest Infection (Infections and infestations) | 0 (0) | 4 (4)
Cryptococcal Meningitis (Infections and infestations) | 1 (1) | 1 (1)
Diarrhoea Cryptosporidial (Infections and infestations) | 1 (1) | 0 (0)
Disseminated Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 3 (3) | 0 (0)
Hidradenitis Suppurativa (Infections and infestations) | 1 (1) | 0 (0)
Joint Infection (Infections and infestations) | 1 (1) | 0 (0)
Lobar Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 4 (4) | 1 (1)
Meningitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic Inflammatory Disease (Infections and infestations) | 1 (1) | 0 (0)
Perineal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pneumocystis Carnii Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia (Infections and infestations) | 6 (6) | 4 (4)
Pulmonary Tuberculosis (Infections and infestations) | 3 (3) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 4 (4) | 0 (0)
Tuberculosis Pleurisy (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis Meningitis (Infections and infestations) | 0 (0) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 0 (0)
Wound Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Chemical Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Motor Vehicle Accident (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Smoke Inhalation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft Tissue Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Stab Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 1 (1) | 2 (2)
ALT Increased (Injury, poisoning and procedural complications) | 7 (9) | 11 (12)
AST Increased (Injury, poisoning and procedural complications) | 5 (5) | 10 (11)
GGT Increased (Investigations) | 7 (8) | 6 (6)
Lipase Increased (Investigations) | 1 (1) | 2 (3)
Loss of Weight (Investigations) | 1 (1) | 1 (1)
Lactate Increased (Investigations) | 0 (0) | 2 (2)
Creatinine Increased (Investigations) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperlactataemia (Metabolism and nutrition disorders) | 3 (3) | 17 (17)
Insulin Dependent Diabetic (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic acidosis (Metabolism and nutrition disorders) | 5 (5) | 9 (9)
Lipodystrophy (Metabolism and nutrition disorders) | 0 (0) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Karposi's Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1)
Left Side Paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Mental Retardation (Nervous system disorders) | 0 (0) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral Neuropathy NOS (Nervous system disorders) | 0 (0) | 1 (1)
Antepartum Haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abruptio Plancentae (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Fetal Death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Hellp Syndrome (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Incomplete Abortion (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Normal Delivery (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Acute Renal Failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Bartholin's Cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal Bleeding (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Parasuicide (Psychiatric disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bullous Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Drug Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Eczema Weeping (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrheic Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Stevens Johnson Syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Assault (Social circumstances) | 2 (2) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Collapse Cardiovascular (Vascular disorders) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 2 (2)
Gangrene (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (4) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Antiretroviral Therapy Monitored by Medical Officer (N=408) | Antiretroviral Therapy Managed by Primary Health Care Nurse (N=404)
Neutropenia (Blood and lymphatic system disorders) | 27 (34) | 17 (22)
GGT increased (Investigations) | 29 (36) | 15 (20) — Gamma Glutamyl Transferase
Hyperlactatemia (Metabolism and nutrition disorders) | 71 (79) | 43 (44)
Lipodystrophy (Skin and subcutaneous tissue disorders) | 39 (40) | 34 (35)
Peripheral Neuropathy (Nervous system disorders) | 28 (29) | 10 (10)

LIMITATIONS AND CAVEATS:
The study design did not address nurse-initiated ART because the prescription of ART in South Africa is restricted to doctors. We noted a high rate of loss to follow-up, but this rate was similar to other resource-constrained settings.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes